CLINICAL TRIAL: NCT07280013
Title: A Phase 1B, Open-label, Multicenter Study to Evaluate the Safety and Preliminary Efficacy of Cemsidomide in Combination With Elranatamab in Relapsed/Refractory Multiple Myeloma Subjects
Brief Title: A Study to Learn About the Effects of Cemsidomide in Combination With Elranatamab in Relapsed/Refractory Multiple Myeloma Subjects
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: C4 Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CFT7455-1102
Record Dates: First submitted 2025-12-01; First posted 2025-12-12 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma (MM)
Keywords: multiple myeloma, cemsidomide, CFT7455, elranatamab, PF-06863135, relapsed, refractory, RRMM, BCMA, bispecific antibody, BiTE, TCE, ELREXFIO
MeSH Terms: conditions — Multiple Myeloma; Recurrence; Bites and Stings

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Non-randomized cemsidomide (tablet) plus elranatamab (subcutaneous injection) (Experimental)
  Interventions: Drug: Cemsidomide; Biological: Elranatamab

INTERVENTIONS:
Drug: Cemsidomide — IKZF1/3 degrader
Biological: Elranatamab — • BCMA-CD3 bispecific antibody
  Other Names: o PF-06863135 o ELREXFIO

SUMMARY:
The main purpose of the study is to understand the safety and tolerability of cemsidomide when given along with elranatamab in subjects with relapsed or refractory multiple myeloma.

The first part of the study will evaluate different dose levels of cemsidomide in combination with elranatamab in a limited number of subjects. Approximately 3 different dose levels of cemsidomide in combination with elranatamab may be explored. Once a dose level is determined safe, additional subjects may be enrolled through expansion of the dose level. This expansion will provide further exploration of the safety and evaluation of preliminary antimyeloma activity.

Cemsidomide will be taken orally each cycle for 14 days on/14 days off (1 cycle=28 days). Elranatamab will be administered by subcutaneous injection twice a month. Dexamethasone will be administered weekly until a confirmed response but no longer than 4 cycles.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of multiple myeloma as defined by IMWG criteria
* Measurable disease based on IMWG criteria
* Received 1-4 prior lines of therapy for multiple myeloma, consisting of at least 1 immunomodulatory drug (i.e., IKZF 1/3 degrader)
* ECOG performance status 0-2

Exclusion Criteria:

* Smoldering multiple myeloma, POEMS Syndrome, systemic light chain amyloidosis, MDS
* Stem cell transplant within 12 weeks prior to enrollment or active graft vs host disease
* Participants with any active, uncontrolled bacterial, fungal, or viral infection
* Prior treatment with a BCMA-directed TCE or BCMA-directed CAR-T therapy
* Administration with an investigational product within 30 days preceding the first dose of study intervention
* Inability or difficulty swallowing tablets, malabsorption syndrome, or any disease or medical condition significantly affecting gastrointestinal function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of cemsidomide in combination with elranatamab | Cycle 1 approximately 28 days
  Dose limiting toxicity rate
Safety and tolerability of cemsidomide in combination with elranatamab | Baseline through 30 days after discontinuation of study treatment
  Frequency and severity of AEs

SECONDARY OUTCOMES:
Assess antimyeloma activity | Approximately 2 years
  Objective Response Rate (ORR) per IMWG criteria
Evaluate the PK of cemsidomide and elranatamab | Approximately 4 months
  Pre and post dose concentrations of cemsidomide
Evaluate the PK of cemsidomide and elranatamab | Approximately 2 years
  Pre dose concentrations of elranatamab
Assess the immunogenicity of elranatamab | Approximately 2 years
  Percent of participants with positive anti-drug antibodies to elranatamab

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - UCLA Health, Jonsson Comprehensive Cancer Center, Santa Monica, California
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - Norton Cancer Institute St. Matthews, Louisville, Kentucky
  - University of Maryland Greenbaum Comprehensive Cancer Center, Baltimore, Maryland
  - START Midwest, Grand Rapids, Michigan
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke Cancer Center, Durham, North Carolina
  - Tennessee Oncology, Nashville, Tennessee
  - Houston Methodist Hospital, Houston, Texas
  - Huntsman Cancer Institute, University of Utah, Salt Lake City, Utah
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No